CLINICAL TRIAL: NCT01331343
Title: The Guard Control Trial - Randomized, Controlled, Muti-centric, Clinical Study to Assess Whether Type 1 Diabetic Patients in Poor Glycemic Control Can Improve Using the Real-time Values of the Guardian RT Versus Conventional Self-Monitoring Blood Glucose
Brief Title: Effectiveness Study of the Guardian RT in Type 1 Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Severine Liabat, Medtronic Internationtal Trading Sarl
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU007_022004
Record Dates: First submitted 2011-04-05; First posted 2011-04-08 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Glycemic Control; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Guardian RT Telemetered Glucose Monitoring System

SUMMARY:
The purpose of this study is to determine whether Type 1 diabetic patients using the Guardian RT glucose sensor can improve glycemic control over a 12-week period, compared to patients using self-monitoring blood glucose testing (SMBG) alone.

DETAILED DESCRIPTION:
The long-term benefit of tight glycemic control in diabetics is well documented. HbA1c generally assesses the average/long term quality of glycemic control. On a daily basis, patients assess their glycemic control through finger stick measurements (SMBG), which allows them to adjust their therapy. A device which would provide a patient with a real-time glucose value, as well as high and low alerts, could aid the patient in knowing when to perform confirmatory SMBG tests and intervene so that dangerous glycemic excursions may occur less frequently.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for at least 12 months
* HbA1c must be 8.1% or above at study entry
* Intensive Insulin Therapy 3 months prior to study entry

Exclusion Criteria:

* Impaired hearing or vision (must see screens and hear alarms)
* Unable to comply with protocol
* Chronic debilitating or psychiatric disturbances

Ages: 8 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Difference in Change in A1c (%) between continuous use of CGM and control | 12 weeks

SECONDARY OUTCOMES:
Difference in change in A1c (%) between biweekly use of CGM and control | 12 weeks
Difference in change in A1c (%) between biweekly use of CGM and continuous use of CGM | 12 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- France (2):
  - Hospital Sud Francilien, Corbeil-Essonnes
  - CH Robert Debre, Paris
- Klinik fur Allgemeine Charite, Berlin, Germany
- Schneider Children Centre, Petah Tikva, Israel
- U.O. Medicina Generale, Milan, Italy
- University Children's Hospital, Ljubljana, Slovenia
- Huddinge University Hospital, Huddinge, Sweden
- Royal Bournemouth Hospital, Dorset, United Kingdom